CLINICAL TRIAL: NCT03800940
Title: Trans-drain Occlusion for Postoperative Pancreatic Fistula- A Double Blind Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201809040RIND
Record Dates: First submitted 2019-01-02; First posted 2019-01-11 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Pancreatic Fistula
MeSH Terms: conditions — Pancreatic Fistula

STUDY DESIGN:
Intervention Model Description: Enrolled patients will be randomly assigned in a 2:1 ratio to receive trans-drain occlusion followed by gradual drain withdrawal or gradual drain withdrawal.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fistulography and trans-drain occlusion (Experimental): Fistulography is performed to assess the condition of the fistula, and trans-drain occlusion is performed by injecting glue (NBCA and Lipiodol) through the drain to occlude the tract.
  Interventions: Procedure: Fistulography and trans-drain occlusion
- Fistulography (Sham Comparator): Fistulography is performed to assess the condition of the fistula, without trains-drain occlusion.
  Interventions: Procedure: Fistulography

INTERVENTIONS:
Procedure: Fistulography and trans-drain occlusion — 1. Fistulography: an 18G needle is inserted into the tube and diluted contrast medium is slowly injected into the tube.
  2. Trans-drain occlusion: a 0.035-inch guidewire is inserted via the puncture needle. The drain tube is removed, cut at 4 cm proximal to the skin fixation site, and preserved for reinsertion. After inserting a 40cm 5Fr KMP catheter over the guidewire, the guidewire is removed. Afte rinsing the KMP catheter with 3ml 5% glucose water, withdraw the catheter and simultaneously inject glue (33%, 1:2, 0.5ml of NBCA + 1ml Lipiodol) into the catheter until the proximal 5cm of the catheter remains inside the tract. The guidewire is re-inserted through the catheter, and then the original drain tube is re-inserted over the guidewire. The guidewire is removed and the drain is fixed.
  Arms: Fistulography and trans-drain occlusion
Procedure: Fistulography — Fistulography: an 18G needle is inserted into the tube and diluted contrast medium is slowly injected into the tube.
  Arms: Fistulography

SUMMARY:
This is a multicenter, investigator initiated, prospective, superiority, parallel-group, randomized, double-blinded trial that aims to compare the efficacy and safety of trans-drain occlusion followed by gradual withdrawal of drain versus gradual withdrawal of drain alone for postoperative pancreatic fistula (POPF) that persists for longer than 21 days.

DETAILED DESCRIPTION:
The most common major complication after pancreatic resection is postoperative pancreatic fistula (POPF), which is defined as a drain output of any measurable volume of fluid on and after postoperative day 3 with an amylase content > 3 times the upper limit of normal serum level. Gradual withdrawal of surgically placed drains in patients who are clinically stable and tolerate a diet is generally adopted to hasten closure of POPF. For high-output fistulas (> 150-200 mL of amylase-rich fluid per day), patients are initially managed with fasting and enteral or parenteral nutrition. If fistula output decreases substantially with these measures and the patient remains clinically well, drain withdrawal is initiated and oral intake is slowly restarted. If the patient remains well despite high fistula output, drains are slowly withdrawn in an attempt to decrease the output and close the fistula. When the output decrease to less than 10 mL per day, the drains are removed.

However, the current standard practice of gradual drain withdrawal is time consuming. Although clinically stable can be discharged with the drain, the drainage tube often remains in place for a prolonged period, with patient discomfort and increased medical cost. In a pilot study by the investigators, 32.5% (37/114) of POPF patients required drainage for longer than 21 days. Besides, there is also considerable risk of recurrent fluid collection along the drain tube tract after drain removal.

The investigators' experience has shown that trans-drain occlusion of the drain tract achieves fistula closure, enabling immediate removal of the drain. In a pilot study, 20 patients underwent trans-catheter occlusion for POPFs that persisted for more than 3 weeks after placement of drainage tubes. No subjective symptoms or abnormalities in blood tests were noted in 17 patients after the procedure. Three patients had abdominal pain without signs of infection, and the pain spontaneously subsided after conservative treatment. POPF healed immediately after occlusion in all of the 20 patients without recurrence during follow-up. This multicenter, investigator initiated, prospective, superiority, parallel-group, randomized, double-blinded trial aims to compare the efficacy and safety of trans-drain occlusion followed by gradual withdrawal of drain versus gradual withdrawal of drain alone for POPF that persists for longer than 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo pancreatectomy (including pancreatoduodenectomy with or without pylorus preservation, distal pancreatectomy, and central pancreatectomy) and develop POPF that persists for 3 weeks after its occurrence.
* With POPF that persists for 3 weeks after occurrence

Exclusion Criteria:

* Younger than 20 years of age
* Active infection not adequately controlled [body temperature ≧38.5℃ and/or eukocytosis (WBC count >15,000 /uL)/leukopenia (WBC count <4,000 /uL)], have residual intra-abdominal fluid collection (largest diameter > 4cm) despite tube drainage on CT scan (with or without contrast, performed when the patient meet inclusion criteria).
* Current or history of severe heart, lung, kidney, or liver failure
* Karnofsky Performance Score <60
* Pregnant or lactating
* Have received somatostatin or its analogue in the index admission
* Decline to participate

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2022-11-27 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Days to fistula closure | The date of fistula closure is the date on which the drain is removed after an output of ≦ 10 mL during 48 hours, without recurrence of fistula within the next 3 months
  Days from the randomly allocated treatment to fistula closure

SECONDARY OUTCOMES:
30-day fistula closure rate | From enrollment to 4 months after fistula occurrence
  Proportion of patients in whom the drain can be removed by 30 days after occurrence of fistula, without recurrence within the next 3 months
Rate of persistent or recurrent POPF after initial drain removal | From drain removal to 3 months after drain removal or recurrence of fistula, whichever occurs first
  Proportion of patients with fluid collection on follow-up CT, which is to be performed at 3 months after removal of drain or when recurrence of fistula is suspected clinically.
Length of hospital stay after the assigned treatment | From treatment to discharge from the index admission, an average of 2 weeks
  Days from the assigned treatment to discharge
Hospital costs after the assigned treatment | From treatment to discharge from the index admission, an average of 2 weeks
  Costs from the assigned treatment to discharge
Rate of fistula-related complications | From occurrence of fistula to 3 months after drain removal
  Proportion of patients who develop fever/infection, ileus, postpancreatectomy hemorrhage from the assigned treatment to end of follow-up.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From treatment to discharge from the index admission, an average of 2 weeks
  Fever/infection or pain that develops within 48 hours after the allocated treatment, or any adverse events judged to be related to the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Wen Tien, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schlitt HJ, Schmidt U, Simunec D, Jager M, Aselmann H, Neipp M, Piso P. Morbidity and mortality associated with pancreatogastrostomy and pancreatojejunostomy following partial pancreatoduodenectomy. Br J Surg. 2002 Oct;89(10):1245-51. doi: 10.1046/j.1365-2168.2002.02202.x. PMID 12296891
- [Background] Balcom JH 4th, Rattner DW, Warshaw AL, Chang Y, Fernandez-del Castillo C. Ten-year experience with 733 pancreatic resections: changing indications, older patients, and decreasing length of hospitalization. Arch Surg. 2001 Apr;136(4):391-8. doi: 10.1001/archsurg.136.4.391. PMID 11296108
- [Background] Yeo CJ, Cameron JL, Sohn TA, Lillemoe KD, Pitt HA, Talamini MA, Hruban RH, Ord SE, Sauter PK, Coleman J, Zahurak ML, Grochow LB, Abrams RA. Six hundred fifty consecutive pancreaticoduodenectomies in the 1990s: pathology, complications, and outcomes. Ann Surg. 1997 Sep;226(3):248-57; discussion 257-60. doi: 10.1097/00000658-199709000-00004. PMID 9339931
- [Background] Bassi C, Marchegiani G, Dervenis C, Sarr M, Abu Hilal M, Adham M, Allen P, Andersson R, Asbun HJ, Besselink MG, Conlon K, Del Chiaro M, Falconi M, Fernandez-Cruz L, Fernandez-Del Castillo C, Fingerhut A, Friess H, Gouma DJ, Hackert T, Izbicki J, Lillemoe KD, Neoptolemos JP, Olah A, Schulick R, Shrikhande SV, Takada T, Takaori K, Traverso W, Vollmer CM, Wolfgang CL, Yeo CJ, Salvia R, Buchler M; International Study Group on Pancreatic Surgery (ISGPS). The 2016 update of the International Study Group (ISGPS) definition and grading of postoperative pancreatic fistula: 11 Years After. Surgery. 2017 Mar;161(3):584-591. doi: 10.1016/j.surg.2016.11.014. Epub 2016 Dec 28. PMID 28040257
- [Background] Bassi C, Dervenis C, Butturini G, Fingerhut A, Yeo C, Izbicki J, Neoptolemos J, Sarr M, Traverso W, Buchler M; International Study Group on Pancreatic Fistula Definition. Postoperative pancreatic fistula: an international study group (ISGPF) definition. Surgery. 2005 Jul;138(1):8-13. doi: 10.1016/j.surg.2005.05.001. PMID 16003309
- [Background] Roberts KJ, Sutcliffe RP, Marudanayagam R, Hodson J, Isaac J, Muiesan P, Navarro A, Patel K, Jah A, Napetti S, Adair A, Lazaridis S, Prachalias A, Shingler G, Al-Sarireh B, Storey R, Smith AM, Shah N, Fusai G, Ahmed J, Abu Hilal M, Mirza DF. Scoring System to Predict Pancreatic Fistula After Pancreaticoduodenectomy: A UK Multicenter Study. Ann Surg. 2015 Jun;261(6):1191-7. doi: 10.1097/SLA.0000000000000997. PMID 25371115
- [Background] El Nakeeb A, Salah T, Sultan A, El Hemaly M, Askr W, Ezzat H, Hamdy E, Atef E, El Hanafy E, El-Geidie A, Abdel Wahab M, Abdallah T. Pancreatic anastomotic leakage after pancreaticoduodenectomy. Risk factors, clinical predictors, and management (single center experience). World J Surg. 2013 Jun;37(6):1405-18. doi: 10.1007/s00268-013-1998-5. PMID 23494109
- [Background] Veillette G, Dominguez I, Ferrone C, Thayer SP, McGrath D, Warshaw AL, Fernandez-del Castillo C. Implications and management of pancreatic fistulas following pancreaticoduodenectomy: the Massachusetts General Hospital experience. Arch Surg. 2008 May;143(5):476-81. doi: 10.1001/archsurg.143.5.476. PMID 18490557
- [Background] McMillan MT, Soi S, Asbun HJ, Ball CG, Bassi C, Beane JD, Behrman SW, Berger AC, Bloomston M, Callery MP, Christein JD, Dixon E, Drebin JA, Castillo CF, Fisher WE, Fong ZV, House MG, Hughes SJ, Kent TS, Kunstman JW, Malleo G, Miller BC, Salem RR, Soares K, Valero V, Wolfgang CL, Vollmer CM Jr. Risk-adjusted Outcomes of Clinically Relevant Pancreatic Fistula Following Pancreatoduodenectomy: A Model for Performance Evaluation. Ann Surg. 2016 Aug;264(2):344-52. doi: 10.1097/SLA.0000000000001537. PMID 26727086
- [Background] Diener MK, Seiler CM, Rossion I, Kleeff J, Glanemann M, Butturini G, Tomazic A, Bruns CJ, Busch OR, Farkas S, Belyaev O, Neoptolemos JP, Halloran C, Keck T, Niedergethmann M, Gellert K, Witzigmann H, Kollmar O, Langer P, Steger U, Neudecker J, Berrevoet F, Ganzera S, Heiss MM, Luntz SP, Bruckner T, Kieser M, Buchler MW. Efficacy of stapler versus hand-sewn closure after distal pancreatectomy (DISPACT): a randomised, controlled multicentre trial. Lancet. 2011 Apr 30;377(9776):1514-22. doi: 10.1016/S0140-6736(11)60237-7. PMID 21529927
- [Background] Tjaden C, Hinz U, Hassenpflug M, Fritz F, Fritz S, Grenacher L, Buchler MW, Hackert T. Fluid collection after distal pancreatectomy: a frequent finding. HPB (Oxford). 2016 Jan;18(1):35-40. doi: 10.1016/j.hpb.2015.10.006. Epub 2015 Nov 18. PMID 26776849

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/40/NCT03800940/Prot_SAP_000.pdf